CLINICAL TRIAL: NCT00845884
Title: A Phase I/II Study Evaluating the Combination of Weekly Docetaxel and Cisplatin Together With Capecitabine and Bevacizumab in Patients With Advanced Gastric Cancer
Brief Title: Phase I/II Study of Weekly Docetaxel and Cisplatin Together With Capecitabine and Bevacizumab in Advanced Gastric Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: Baruch Brenner, MD, Davidoff Cancer Center, Rabin Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AVDCF-2008
Record Dates: First submitted 2009-02-16; First posted 2009-02-18 (Estimated); Last update posted 2009-02-18 (Estimated); Status verified 2009-02

CONDITIONS: Advanced Gastric Cancer
Keywords: Gastric; Cancer; Advanced; Docetaxel; Cisplatin; Capecitabine; Bevacizumab
MeSH Terms: conditions — Neoplasms | interventions — Docetaxel; Cisplatin; Capecitabine; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AVDCF (Experimental): Drug: Docetaxel, Cisplatin, Capecitabine, Bevacizumab
  Interventions: Drug: Docetaxel, Cisplatin, Capecitabine, Bevacizumab

INTERVENTIONS:
Drug: Docetaxel, Cisplatin, Capecitabine, Bevacizumab — * Docetaxel 30-35 mg/m2 IV, on Days 1 and 8, Q:21 days.
  * Cisplatin 30-35 mg/m2 IV, on Days 1 and 8, Q:21 days.
  * Capecitabine 1,600 mg/m2/d PO, divided into two daily doses, on Days 1-14, Q:21 days.
  * Bevacizumab 7.5 mg/kg IV, on Day 1, Q:21 days.
  Other Names: Taxotere (Docetaxel); Cisplatin; Xeloda (Capecitabine); Avastin (Bevacizumab

SUMMARY:
In spite of multiple attempts to improve the efficacy of first-line chemotherapy in advanced gastric cancer, the progress that has been achieved so far is rather limited, and many investigators are exploring newer regimens.A combination of decetaxel (Taxotere) with Cisplatin and 5-fluorouracil (5FU) is considered one of the most effective regimens in this disease. However, it is associated with significant toxicity which avoided its general adaptation by the medical community. The current study is exploring a newer way to administer these three drugs, hopefully making the regimen more comfortable, less toxic and maybe even more effective. We will do this by changing the dose and timing of Taxotere and Cisplating, by replacing protracted infusion of 5FU with tablets of Capecitabine (Xeloda) and by adding the anti-angiogenic drug, Bevacizumab (Avastin), which had shown encouraging results in this disease.

ELIGIBILITY:
Inclusion Criteria:

1. Patients above 18 years of age at the time of enrollment.
2. Histologically confirmed previously untreated metastatic or unresectable adenocarcinoma of the stomach.
3. Patients must have at least one measurable lesion (measuring >10mm in standard CT or >5mm in spiral CT).
4. Adequate organ function.
5. Life expectancy of at least three months.
6. Patients must have an ECOG Performance Status of 0 or 1.
7. Signed written informed consent to participate in the study.

Exclusion Criteria:

1. Participation in an investigational trial within 30 days of the screening visit.
2. Known allergy or any other adverse reaction to any of the study drugs or to any related compound.
3. Prior anti-angiogenic treatment, chemotherapy or radiotherapy for advanced disease. Patients will be eligible if they had received adjuvant chemotherapy or radiotherapy more than 12 months prior to enrollment.
4. Prior treatment with drugs included in the investigational regimen. Prior use of 5-fluorouracil in the adjuvant setting is allowed.
5. Significant bleeding by the primary tumor (in unoperated patients).
6. Clinically significant (i.e. active) cardiovascular disease. This includes, but is not limited to, the following examples:

   * Cerebrovascular accidents (up to 6 months prior to randomization)
   * Myocardial infarction (up to 1 year prior to randomization).
   * Uncontrolled hypertension (above 150/100 mmHg) while receiving chronic medication
   * Unstable angina
   * New York Heart Association (NYHA) Grade II or greater congestive heart failure.
   * Serious cardiac arrhythmia requiring medication.
   * Clinically significant ECG findings. Patients who suffer from serious cardiac arrhythmia requiring medication can enter the study only if they are considered to be in a stable condition regarding both the arrhythmia and their medication. Patients with pacemakers are allowed to enter the study only if they are considered as being in a stable condition. In case of doubt, the investigator should obtain a consultation with a local cardiologist.
7. Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to study treatment start, not fully healed wounds, or anticipation of the need for major surgical procedure during the course of the study.
8. Severe co-morbid conditions including uncontrolled diabetes or hypertension, cerebral vascular disease or uncontrolled infection.
9. Fertile subjects who are not willing to use an acceptable method of contraception during the treatment period and for 28 days following completion of treatment
10. For women of child-bearing potential: a positive pregnancy test at screening or breast-feeding.
11. History of prior malignancy (other than non-melanoma skin cancer, in-situ cervical cancer, or superficial transitional cell bladder cancer) in the last 5 years prior to enrollment.
12. Clinically significant hearing loss.
13. Patients with a history of seizure disorder who are receiving phenytoin, phenobarbital, or other antiepileptic medication.
14. Known peripheral neuropathy of CTCAE v 3.0 Grade 1 or more.
15. Organ allografts requiring immunosuppressive therapy.
16. Serious, non-healing wound, ulcer, or bone fracture.

    -

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Estimated)
Dates: Start 2009-02; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
response rate | 2/2009-12/2012

SECONDARY OUTCOMES:
Safety, PFS, overall survival | 2/2009-12/2012

CONTACTS AND LOCATIONS:
Overall Officials: Baruch Brenner, MD, Principal Investigator — Davidoff Cancer Center, Rabin Medical Center
Locations (1):
- Davidoff Cancer Center, Rabin Medical Center, Petah Tikva, Israel

REFERENCES:
- [Derived] Brenner B, Sarfaty M, Purim O, Kundel Y, Amit L, Abramovich A, Sadeh Gonik U, Idelevich E, Gordon N, Medalia G, Sulkes A. A Phase Ib/II Study Evaluating the Combination of Weekly Docetaxel and Cisplatin Together with Capecitabine and Bevacizumab in Patients with Advanced Esophago-Gastric Cancer. PLoS One. 2016 Jul 8;11(7):e0157548. doi: 10.1371/journal.pone.0157548. eCollection 2016. PMID 27390847